CLINICAL TRIAL: NCT07342374
Title: Optimising Bolus Tracking Technique by Repositioning the Region of Interest (ROI) at the Superior Vena Cava and Reducing Contrast Media Volume in Computed Tomography Pulmonary Angiography (CTPA)
Brief Title: Repositioning the Bolus Tracking ROI to the Superior Vena Cava in CTPA Facilitates Contrast Volume Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Queen Elizabeth, Malaysia (Other Government)
Collaborators: Universiti Sultan Zainal Abidin (Other)
Responsible Party: Principal Investigator, MOHD ARI-NADZAHARI BIN ABD RAHMAN, Diagnostic Radiographer, Hospital Queen Elizabeth, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NMRR-20-699-54086 (IIR)
Record Dates: First submitted 2026-01-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Artery Embolism; Pulmonary Embolism (PE)
Keywords: Pulmonary Embolism; Computed Tomography Pulmonary Angiography; Contrast Media; Bolus Tracking; Superior Vena Cava; Image Quality; Low-volume Protocol
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Intervention Model Description: This study uses a four-arm parallel assignment to compare two primary factors: the anatomical location of the bolus-tracking region of interest (ROI) and the volume of contrast media administered. Participants are randomized into one of four distinct protocol groups (Groups A, B, C, or D) to evaluate image quality and opacification differences across the various combinations of ROI placement (Pulmonary Trunk vs. Superior Vena Cava) and contrast volume (50 ml vs. 30 ml).
Who Masked: Outcomes Assessor
Masking Description: Three senior radiologists served as blinded outcomes assessors for this study. These assessors were blinded to all protocol details, including the anatomical location of the bolus-tracking region of interest (ROI) and the volume of contrast media administered for each participant. The CTPA images were anonymized and presented to the assessors in a randomized order to ensure objective qualitative evaluation of image quality using the 5-point Likert scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: PT-ROI, 50 ml (Control) (Active Comparator): Standard CTPA protocol using the bolus tracking technique with the monitoring region of interest (ROI) placed at the pulmonary trunk (PT) and 50 ml of contrast media.
  Interventions: Diagnostic Test: Optimized CTPA Protocol
- Group B: PT-ROI, 30 ml (Experimental): Modified CTPA protocol using the bolus tracking technique with the monitoring ROI at the pulmonary trunk (PT) and a reduced contrast volume of 30 ml.
  Interventions: Diagnostic Test: Optimized CTPA Protocol
- Group C: SVC-ROI, 50 ml (Experimental): Modified CTPA protocol using the bolus tracking technique with the monitoring ROI repositioned upstream to the superior vena cava (SVC) and 50 ml of contrast media.
  Interventions: Diagnostic Test: Optimized CTPA Protocol
- Group D: SVC-ROI, 30 ml (Experimental): Modified CTPA protocol using the bolus tracking technique with the monitoring ROI repositioned upstream to the superior vena cava (SVC) and a reduced contrast volume of 30 ml.
  Interventions: Diagnostic Test: Optimized CTPA Protocol

INTERVENTIONS:
Diagnostic Test: Optimized CTPA Protocol — CTPA scans are performed on a 128-slice CT scanner using the bolus tracking technique. Non-ionic contrast medium (370 mgI/ml) is administered at a rate of 4 ml/s, followed by a 20 ml saline flush. The diagnostic scan is automatically triggered when enhancement in the monitoring region of interest (ROI) reaches a threshold of 100 HU, with a fixed transit delay time (TDT) of 5 seconds.

SUMMARY:
This randomized controlled trial evaluates a protocol optimization for Computed Tomography Pulmonary Angiography (CTPA). The study investigates the impact of repositioning the bolus-tracking region-of-interest (ROI) from the standard pulmonary trunk (PT) to the superior vena cava (SVC). The goal is to compensate for the CT scanner's inherent transit delay time (TDT) to better align the scan with the peak arterial phase. By optimizing this timing, the study assesses whether contrast media volume can be safely reduced by 40% (from 50 ml to 30 ml) while maintaining diagnostic image quality and preventing venous contamination.

DETAILED DESCRIPTION:
Background and Rationale: Computed Tomography Pulmonary Angiography (CTPA) is the gold standard for diagnosing pulmonary embolism (PE). However, standard bolus tracking (BT) protocols that place the monitoring region-of-interest (ROI) on the main pulmonary trunk (PT) often face challenges due to the system's inherent Transit Delay Time (TDT). This delay, typically 5 seconds, can cause the diagnostic scan window to overlap with the venous phase, leading to suboptimal arterial opacification and venous contamination. This study proposes repositioning the monitoring ROI upstream to the superior vena cava (SVC) to utilize the TDT as transit time for the bolus, thereby aligning the scan window with the peak arterial phase.

Study Objectives: The primary objective is to evaluate the effect of SVC ROI repositioning on diagnostic image quality while investigating the feasibility of reducing contrast media (CM) volume by 40% (from 50 ml to 30 ml).

Methodology: This is a single-center, prospective, randomized controlled trial involving 72 adult patients. Participants are randomized into four protocol groups:

Group A (Control): ROI at PT, 50 ml contrast media. Group B: ROI at PT, 30 ml contrast media. Group C: ROI at SVC, 50 ml contrast media. Group D: ROI at SVC, 30 ml contrast media.

Protocol Details:

* Contrast Administration: Non-ionic contrast medium (370 mgI/ml) is injected at a rate of 4 ml/s, followed by a 20 ml saline flush.
* Bolus Tracking: An elliptical ROI is placed either on the PT (above the carina) or SVC depending on the group assignment.
* Triggering: The diagnostic scan is automatically initiated when enhancement reaches a threshold of 100 HU. The TDT is set to a fixed 5 seconds.
* Assessment: Diagnostic quality is assessed quantitatively by calculating arterial-venous enhancement differences (HU) and qualitatively via a 5-point Likert scale by three blinded radiologists.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for a Computed Tomography Pulmonary Angiography (CTPA) examination.
* Provision of written informed consent by the subject, guardian, or medical specialist.
* Patients with an upper extremity intravenous (IV) line using a 16-20 gauge cannula.
* Patients with a stable heart rate between 60 and 120 beats per minute (bpm).

Exclusion Criteria:

* Pregnancy, breastfeeding, or use of non-reliable methods of contraception.
* Patients with impaired renal function, including acute kidney injury or chronic kidney disease (CKD) with an eGFR less than 30 mL/min/1.73m².
* Patients with a lower extremity IV line, as this bypasses the Superior Vena Cava (SVC) and results in bolus tracking technique failure.
* Patients with a heart rate lower than 60 bpm or higher than 120 bpm.
* Patients with a cannula size of 22g or smaller, as it cannot accommodate the high flow rate (4 mL/s) required by the power injector.
* Patients with severe cardiac impairment or congenital heart disease.
* Patients with a Body Mass Index (BMI) exceeding 35 kg/m², as severe obesity causes beam hardening effects that degrade image quality.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Mean Difference in Hounsfield Unit (HU) Attenuation Between Pulmonary Artery and Pulmonary Vein | At the time of post-procedural image analysis (approximately 48 hours after CTPA scan completion).
  This quantitative measurement assesses the degree of arterial opacification relative to venous contamination by calculating the difference in Hounsfield Units (HU). It is calculated by subtracting the mean HU value of the pulmonary vein from the mean HU value of the pulmonary artery at the same anatomical level. A larger positive difference indicates superior arterial enhancement with minimal venous contamination.

SECONDARY OUTCOMES:
Qualitative Image Quality Score using a 5-point Likert Scale | Within 1 month following the CTPA scan.
  Qualitative assessment of CTPA images performed by three blinded senior radiologists using a 5-point Likert scale (1 = Unacceptable, 2 = Sub-optimal, 3 = Acceptable, 4 = Good, 5 = Excellent). The score evaluates overall arterial enhancement, presence of artifacts, and diagnostic adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Kamarul Amin. bin Abdullah @ Abu Bakar., Assoc. Prof. Ts. Dr., Study Chair — Universiti Sultan Zainal Abidin (UniSZA)
Locations (1):
- Hospital Queen Elizabeth, Kota Kinabalu, Sabah, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be kept strictly confidential in accordance with the hospital's privacy policies and the informed consent agreement. To protect participant privacy, only aggregated results and statistical data will be reported in publications.